CLINICAL TRIAL: NCT05842863
Title: Combined Dialectical Behavior Therapy and Digital Cognitive Behavioral Therapy for Insomnia for Adolescents at High Risk for Suicide: A Pilot RCT
Brief Title: Combined Dialectical Behavior Therapy and Digital Cognitive Behavioral Therapy for Insomnia for Adolescents at High Risk for Suicide
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michele Berk, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69003; 1R34MH130634-01A1 (NIH)
Record Dates: First submitted 2023-04-18; First posted 2023-05-06 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Suicide and Self-harm
MeSH Terms: conditions — Suicide; Self-Injurious Behavior | interventions — Dialectical Behavior Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dialectical Behavior Therapy + Cognitive Behavioral Therapy for Insomnia (Experimental)
  Interventions: Behavioral: Dialectical Behavior Therapy; Behavioral: Cognitive Behavioral Therapy for Insomnia
- Dialectical Behavior Therapy Only (Active Comparator)
  Interventions: Behavioral: Dialectical Behavior Therapy

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — Dialectical Behavior Therapy (DBT) is a treatment program that helps teens reduce suicidal and self-harm behaviors by teaching them coping skills for managing negative emotions. DBT includes weekly individual therapy, weekly multifamily skills group, and 24/7 telephone-based skills coaching from the therapist.
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia (CBTI) is a type of counseling that helps people improve sleep by changing their sleep behaviors and thinking about sleep. In CBTI, people learn about sleep regulation, factors that influence quantity and quality of sleep, and specific techniques to optimize sleep. In this study, CBTI will be delivered using a self-guided online program called Firefly.
  Arms: Dialectical Behavior Therapy + Cognitive Behavioral Therapy for Insomnia

SUMMARY:
The proposed research addresses the urgent need to reduce suicide rates among teens. This will be the first study that the investigators know of that will examine the feasibility and preliminary effectiveness of augmenting a suicide-focused treatment (Dialectical Behavior Therapy, [DBT]) with an evidence-based treatment protocol for insomnia (a digital version of Cognitive Behavioral Therapy for Insomnia [CBT-I]). The goal of this clinical trial is to learn providing insomnia treatment in conjunction with suicide-focused treatment leads to greater reductions in suicidality and self-harm than suicide-focused treatment alone.

Participants will be randomly assigned to receive 6 months of DBT plus CBT-I or to DBT alone and will complete research assessments measuring suicidal ideation, self-harm behavior and insomnia symptoms every four weeks over the course of the study, as well as one post-treatment follow-up assessment. Participants will also wear a device on their wrist (like a Fitbit or wristwatch) for 10 days following each assessment to collect data about their sleep.

ELIGIBILITY:
Inclusion Criteria:

1. 12-18 years of age and not yet graduated from high school.
2. Insomnia symptoms, defined as a total score of ≥ 8 on the Insomnia Severity Index .
3. High suicide risk, defined as: >1 lifetime suicide attempt, b) > 3 lifetime SH episodes (with at least 1 in the 12 weeks before baseline screening) and c) elevated SI (≥31 on the SIQ-Jr.).
4. If taking medication for psychiatric disorders or sleep, must be on a stable dose (>2 months).
5. Youth and parent both speak English.
6. At least one family member or responsible adult agrees to participate in assessments and in the DBT multi-family skills group.
7. Youth lives at home.

Exclusion Criteria:

1. Significant current mania or psychosis; life threatening anorexia, or other diagnosis of a severe mental or physical condition requiring treatment specific to that disorder and/or that interferes with participation in assessments or treatment.
2. A history of being diagnosed with an Autism Spectrum Disorder.
3. Has a comorbid untreated sleep apnea or a severe circadian sleep-wake disorder with a habitual bedtime after 3 AM or habitual rise time after 11 AM.
4. Insomnia symptoms are significantly impacted by substance use or withdrawal of psychoactive medications.
5. Has conditions that require caution when implementing CBTI, such as bipolar and seizure disorders.
6. Court-ordered to treatment.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation Questionnaire Junior (SIQ-JR) | Baseline and change from baseline at 4, 8, 12, 16, 20, 24 and 36 weeks after the start of the DBT program.
  The SIQ-JR (Reynolds 1987) is a 15-item self-report questionnaire that assesses suicidal thoughts on a 7-point scale (I never had this thought to almost every day). Scores range from 0 to 90, with a published clinical cut-off score of 31.
Insomnia Severity Index (ISI) | Baseline and change from baseline at 4, 8, 12, 16, 20, 24 and 36 weeks after the start of the DBT program.
  The ISI (Morin, 1993) is a 7-item self-report questionnaire that measures insomnia symptoms on a 4-point scale. Total score ranges from 0-28, with a total score of > 9 being validated as the optimal cutoff for a likely insomnia diagnosis.
Suicide Attempt Self-Injury Interview and Count | Baseline and change from baseline at 4, 8, 12, 16, 20, 24 and 36 weeks after the start of the DBT program.
  Structured clinical interview that measures number, dates, method, intent and lethality of suicide attempts and non-suicidal self-injury episodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Michele Berk, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No